CLINICAL TRIAL: NCT04955730
Title: Randomized Trial of Prolonged Use of Negative Pressure Wound Therapy in Patients Undergoing Surgical Procedures for the Management of Gastrointestinal Malignancies
Brief Title: NPWT in Patients Undergoing Surgical Procedures for Management of GI Malignancies
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MCC-20561
Record Dates: First submitted 2021-06-29; First posted 2021-07-09 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and statisticians will be blinded to treatment randomization. Surgical oncologists will be blinded of treatment randomization until the dressing is applied to the wound.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NPWT - Negative Pressure Wound Therapy (Experimental): Participants will receive Negative Pressure Wound Therapy (NPWT) after surgery and wear the NPWT until postop day 3. NPWT dressing will be removed and a new NPWT will be replaced until Postop day 7, where NPWT dressing will be removed.
  Interventions: Device: Negative Pressure Wound Therapy
- Standard of Care Wound Therapy (No Intervention): Participants will receive standard of care wound therapy after surgery. Postop day 3, dressings will be removed and new sterile dressings will be applied if needed.

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — Negative Pressure Wound Therapy is a single use NPWT that produces a negative pressure at -80 mmHg. Participants will have their fascia and skin closed in the same manner as the control arm participants, and will wear the NPWT dressing for 7 days after surgery.
  Other Names: PICO
  Arms: NPWT - Negative Pressure Wound Therapy

SUMMARY:
This randomized trial will use a Negative Pressure Wound Therapy device or standard wound closure, in participants with gastrointestinal neoplasms, to measure the rate of surgical site infections

ELIGIBILITY:
Inclusion Criteria:

* Scheduled surgical procedure for the management of gastrointestinal cancer
* Scheduled surgical procedure planned for incision that will result in wound >5cm
* Scheduled surgical procedure planned for skin wound that will be closed by primary intention with either: Staples covered by sterile Telfa® and Tegaderm® or Medipore® OR Dermal or subcuticular sutures covered by Octil®
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Scheduled surgical procedure where wound considered dirty
* Scheduled surgical procedure for wound left for closure by secondary intention
* Emergency surgery
* Pregnancy. Pregnancy status is confirmed per protocol the day of surgery in the preoperative space by urine pregnancy test in patient younger than 65 and with intact uterus. Pregnant patient will be excluded from this study
* History or current diagnosis of any medical or psychological condition that in the Investigator's opinion, might interfere with the subject's ability to participate in the study or the inability to obtain informed consent because of psychiatric or complicating medical problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection - Superficial Incisional | 30 days post operation
  Investigators will measure rate of Surgical Site Infection (SSI) of participants who received Superficial Incisions.
Surgical Site Infection - Deep Incisional | 30 days post operation
  Investigators will measure rate of Surgical Site Infection (SSI) of participants who received Deep Incisions.
Surgical Site Infection - Organ/Space Incisional | 30 days post operation
  Investigators will measure rate of Surgical Site Infection (SSI) of participants who received Organ/Space Incisions.

SECONDARY OUTCOMES:
Return to Intended Oncologic Therapy (RIOT) | Up to 12 months after surgery
  Investigators will measure number of participants who returned to their intended oncologic therapy
Time to Initiation of Planned Oncologic Therapy | Up to 12 months after surgery
  Investigators will measure time to initiation planned therapy from the surgery date to initiation date of planned oncologic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Pimiento, MD, Principal Investigator — Moffitt Cancer Center; Daniel Anaya, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinicaltrialssearch?DiseaseSite=&q=20561